CLINICAL TRIAL: NCT02398383
Title: Role of Glucagon in Glucose Control in Cystic Fibrosis Related Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1409014580
Record Dates: First submitted 2015-01-22; First posted 2015-03-25 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis Related Diabetes
MeSH Terms: conditions — Cystic Fibrosis | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CF with Normal Glucose Tolerance (Experimental): Individuals with CF without cystic fibrosis related diabetes
  Interventions: Other: Oral Glucose Tolerance Test; Other: Mixed Meal Tolerance Test; Other: Hypoglycemic Clamp
- Cystic Fibrosis Related Diabetes (Experimental): Individuals with cystic fibrosis and cystic fibrosis related diabetes
  Interventions: Other: Oral Glucose Tolerance Test; Other: Mixed Meal Tolerance Test; Other: Hypoglycemic Clamp
- Control (Active Comparator): Age matched control subjects
  Interventions: Other: Oral Glucose Tolerance Test; Other: Mixed Meal Tolerance Test; Other: Hypoglycemic Clamp

INTERVENTIONS:
Other: Oral Glucose Tolerance Test — Subjects will be instructed to fast after midnight the night prior to the study. Subjects will be admitted to the research unit on the morning of the test for placement of blood-drawing IV for frequent sampling. Patients will drink 1.75 gm/kg glucose (Glucola) to a maximum of 75 gm. Venous samples for glucose and c-peptide will be drawn from the IV at 0, 30, 60, 90 and 120 minutes. Subjects will be instructed to eat at least 75 gm carbohydrates daily in the week prior to this test.
Other: Mixed Meal Tolerance Test — Subjects will be instructed to fast after midnight the night prior to the study. Subjects will be admitted to the research unit on the morning of the test for placement of blood-drawing IV for frequent sampling. Subjects will consume 6 kcal/kg (6 ml/kg) Boost High Protein Nutritional Energy Drink (Mead-Johnson) over five minutes to a maximum of 360 ml. Venous samples for glucose, glucagon, GLP-1, GIP, and c-peptide will be drawn at -10, 0, 15, 30, 60, 90, 120, 150, 180, 210, and 240 minutes.
Other: Hypoglycemic Clamp — All subjects with CF and adult (but not pediatric) controls will undergo one-step hypoglycemic clamp. Subjects will be instructed to fast after midnight the night prior to the study. Subjects will be admitted to the research unit on the morning of the test for placement of blood-drawing IV for frequent sampling and a second IV for infusion of insulin and dextrose.

SUMMARY:
This project is designed to begin to characterize the abnormalities of glucagon secretion in subjects with cystic fibrosis related diabetes along the spectrum of glucose tolerance. Cystic fibrosis patients with normal glucose tolerance as well as cystic fibrosis related diabetes as well as control subjects will undergo an oral glucose tolerance test, mixed meal tolerance test, and one step hypoglycemic clamp. Cystic fibrosis patients will then return 12 months later to undergo repeat mixed meal tolerance test and hypoglycemic clamp test.

DETAILED DESCRIPTION:
This project is designed to begin to characterize the abnormalities of glucagon secretion in subjects with cystic fibrosis related diabetes along the spectrum of glucose tolerance. This will be a descriptive, cross-sectional and longitudinal cohort study in a sample of children and young adults with CF and a continuum of glucose tolerance compared to healthy age-matched controls.

Cystic fibrosis patients with normal glucose tolerance as well as cystic fibrosis related diabetes as well as control subjects will be admitted to the research unit on three separate occasions to undergo an oral glucose tolerance test, mixed meal tolerance test, and one step hypoglycemic clamp. Cystic fibrosis patients will then return 12 months later to undergo repeat mixed meal tolerance test and hypoglycemic clamp test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF by clinical or genetic determination
* Normal glucose tolerance or CFRD
* Subjects routinely taking systemic or inhaled glucocorticoids on stable regimen are eligible

Exclusion Criteria:

* Subjects with active pulmonary infection requiring supplemental doses of corticosteroids
* Use of any oral diabetes medications
* Subjects who are pregnant/lactating
* Subjects with poor compliance with pancreatic enzyme replacement therapy

Control Subjects:

Approximately 10 control subjects who are matched for age, gender, are expected to be enrolled in the study. Non-CF subjects must be >12 years old, in good health and not taking any medications or have any medical problems the doctor feels would prevent the subject from completing the study and have BMI between 15-85% for age and gender. Control subjects whose fasting blood glucose is found to be >110 mg/dL will not be continued in the study.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2015-03; Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Glucagon levels | baseline
  Glucagon levels in response to to a mixed meal stimulus

SECONDARY OUTCOMES:
C-peptide levels | baseline
  C-peptide levels during oral glucose tolerance test and mixed meal tolerance test
C-peptide levels | 12 months
  C-peptide levels during oral glucose tolerance test and mixed meal tolerance test
Epinephrine levels | baseline
  Epinephrine and norepinephrine levels during hypoglycemic clamp
Epinephrine levels | 12 months
  Epinephrine and norepinephrine levels during hypoglycemic clamp
Norepinephrine levels | baseline
  norepinephrine levels during hypoglycemic clamp
Norepinephrine levels | 12 months
  norepinephrine levels during hypoglycemic clamp
Hypoglycemia unawareness scores | Baseline
  Hypoglycemia unawareness scores in subjects during hypoglycemic clamps as measured by the Clarke Hypoglycemia Awareness survey
Hypoglycemia unawareness scores | 12 months
  Hypoglycemia unawareness scores in subjects during hypoglycemic clamps as measured by the Clarke Hypoglycemia Awareness survey
GLP-1 and GIP levels | Baseline
  GLP-1 and GIP levels in response to mixed meal stimulus
GLP-1 and GIP levels | 12 months
  GLP-1 and GIP levels in response to mixed meal stimulus
Glucagon levels | 12 months
  Glucagon levels in response to to a mixed meal stimulus and difference from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bracha Goldsweig, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States